CLINICAL TRIAL: NCT06920433
Title: A Clinical Study Evaluating the Safety and Preliminary Efficacy of Universal Allogeneic CAR T-cell Therapy Targeting CD19 and BCMA in Patients With Relapsed / Refractory Systemic Lupus Erythematosus
Brief Title: UCAR T-cell Therapy Targeting CD19/BCMA in Patients With r/r Systemic Lupus Erythematosus
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Shanghai Xiniao Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Principal Investigator, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH-ZY-01
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: CD19/BCMA CAR T-cells; Universal Allogeneic CAR T-cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCAR T-cell group (Experimental): Universal allogeneic CD19/BCMA CAR T-cells
  Interventions: Biological: UCAR T-cell group

INTERVENTIONS:
Biological: UCAR T-cell group — A single injection of UCAR T-cells, referred to as universal allogeneic anti-CD19/BCMA CAR T-cells

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 18 participants with relapsed or refractory Systemic lupus erythematosus. This study aims to evaluate the safety and efficacy of the treatment with universal CD19/BCMA CAR T-cells.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy of universal CD19/BCMA CAR T-cells in Relapsed or Refractory Systemic lupus erythematosus.

Study intervention consists of a single infusion of universal CAR T-cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

Interim analysis will be performed when participants finish the visit 90 days after CAR T-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Meet the 2019 European League against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for systemic lupus erythematosus; The diagnosis of lupus nephritis was consistent with renal biopsy within 6 months prior to the study, and the histological diagnosis (ISN/RPS2018 LN classification) was active nephritis type III or IV with or without type V. Meet the definition of refractory recurrence: conventional treatment remains ineffective for more than 6 months, or disease activity reappears after remission. Conventional treatment is defined as the use of glucocorticoids, along with one or more of the following immunomodulatory drugs: cyclophosphamide, antimalarial drugs, azathioprine, Mycophenolate Mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics such as rituximab, Beliumab, and Telitacicept.
3. SLEDAI-2000 ≥8；
4. The NIH activity index (AI) of lupus nephritis was >2, and the chronicity index (CI) was increased; Urinary protein: creatinine ratio (UPCR)>1.0g/g, or 24-hour urinary protein >0.5g, with or without active urinary sediment with red blood cell precipitation.
5. Flow cytometry detected positive B cell CD19 or BCMA in the patient's peripheral blood.
6. Functional requirements for major organs are as follows:

   1. The bone marrow function needs to meet: a Neutrophil count ≥ 0.5× 10 ^ 9/L; b. Hemoglobin ≥60g/L: c. Platelets ≥ 20 × 10 ^ 9/L.
   2. Liver function: ALT ≤ 3 × UL; AST ≤ 3×ULN# Total bilirubin ≤ 2.0 ×ULN (excluding Gilbert syndrome, total bilirubin ≤ 3.0 × ULN).
   3. Renal function: creatinine clearance rate (CrCl) ≥ 30 ml/min(Cockcroft/Gault formula, excluding acute CrCl decline caused by the disease itself).
7. ECOG：0-1；
8. Female subjects of childbearing potential and male subjects with partners of childbearing potential must use medically approved contraception or abstinence during the study treatment period and for at least 6 months after the end of the study treatment; Female subjects of childbearing potential must have a negative Human chorionic gonadotropin (HCG) test within 7 days before study enrollment and not be lactating.
9. Willing to participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Subjects with a history of severe drug allergies or allergic tendencies.
2. Presence or suspicion of uncontrolled or treatment-required fungal,bacterial, viral, or other infections.
3. Subjects with central nervous system diseases caused by autoimmune diseases or non-autoimmune diseases (including epilepsy, psychosis, organic brain syndrome, cerebral vascular accidents, encephalitis, central nervous system vasculitis).
4. Subjects with insufficient cardiac function
5. Subjects with congenital immunoglobulin deficiencies
6. History of malignancy within five years
7. Subjects with end-stage renal failure
8. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA titer higher than the upper limit of detection; subjects positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; individuals positive for human immunodeficiency virus (HIV)
9. Subjects with psychiatric disorders and severe cognitive impairments
10. Subjects who had participated in other clinical trials within 3 months prior to enrollment
11. Subjects who have used immunosuppressive agents or biologics with therapeutic effects on the disease within five half-life before enrollment
12. Pregnant women or women planning to conceive
13. Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The number and severity of dose-limiting toxicity (DLT) events | Within 28 Days After UCAR T-cell Infusion
  DLT will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, and the ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells.
The total number, incidence, and severity of AEs | Up to 90 days After UCAR T-cell Infusion
Clinical response | Up to 24 Months After UCAR T-cell Infusion
  SLE：SLE Response Index 4 (SRI-4) LN：Primary effcacy renal response（PERR）

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China